CLINICAL TRIAL: NCT00155766
Title: A Pilot Study for the Immunotherapy of Recurrent Cervical Cancers Using Dendritic Cells (DCs) Pulsed With Human Papillomavirus Type 16 E7 Antigen
Brief Title: Immunotherapy of Recurrent Cervical Cancers Using Dendritic Cells (DCs)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9100205963
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2002-06

CONDITIONS: Cervical Cancer
Keywords: cervical cancer, immunotherapy, DC
MeSH Terms: conditions — Uterine Cervical Neoplasms

INTERVENTIONS:
Biological: HPV16 E7 peptide-pulsed autologous DCs

SUMMARY:
Chemotherapy is the current standard treatment for unresectable recurrent cervical carcinoma after radiotherapy or distant metastasis of cervical carcinoma. The most effective regimens are cisplatin-based chemotherapy. After failure of the cisplatin-based chemotherapy, there is still no treatment that has been proved to be effective.

Human papilloma viruses (HPV) have been consistently implicated in causing cervical cancer especially those high-risk types (HPV 16,18,31,45) have been strongly associated with cervical cancer. HPV 16 was found in more than 50% of cervical cancer tissues. Results from many animal tumor models have indicated that immunization with tumor antigen-pulsed dendritic cells can trigger a long-lasting anti-tumor immune response and significantly inhibit the growth of implanted tumor cells. Recently, many clinical trials have been conducted to evaluate the feasibility and safety of immunizing cancer patients with tumor antigen-pulsed dendritic cells. No severe toxicity has been reported and some patients were shown to respond to the treatment. Based on previous animal and clinical studies by other investigators, we propose to evaluate the potential of immunizing cancer patients with antigen-pulsed autologous dendritic cells as a cancer vaccine to treat for recurrent cervical cancers after failure of cisplatin-based chemotherapy treatment or refusing chemotherapy. In this study, we will generate dendritic cells by culturing patient's autologous PBMC with GM-CSF and IL-4 in vitro. These dendritic cells will be pulsed with synthetic peptides representing the CTL epitopes on HPV Type 16 E7. Antigen-pulsed dendritic cells will be injected into inguinal lymph nodes under the guidance of real-time sonography. Each patient will receive four injections and 12 patients in total will be recruited for this study.

DETAILED DESCRIPTION:
Chemotherapy is the current standard treatment for unresectable recurrent cervical carcinoma after radiotherapy or distant metastasis of cervical carcinoma. The most effective regimens are cisplatin-based chemotherapy. After failure of the cisplatin-based chemotherapy, there is still no treatment that has been proved to be effective.

Human papilloma viruses (HPV) have been consistently implicated in causing cervical cancer especially those high-risk types (HPV 16,18,31,45) have been strongly associated with cervical cancer. HPV 16 was found in more than 50% of cervical cancer tissues. Results from many animal tumor models have indicated that immunization with tumor antigen-pulsed dendritic cells can trigger a long-lasting anti-tumor immune response and significantly inhibit the growth of implanted tumor cells. Recently, many clinical trials have been conducted to evaluate the feasibility and safety of immunizing cancer patients with tumor antigen-pulsed dendritic cells. No severe toxicity has been reported and some patients were shown to respond to the treatment. Based on previous animal and clinical studies by other investigators, we propose to evaluate the potential of immunizing cancer patients with antigen-pulsed autologous dendritic cells as a cancer vaccine to treat for recurrent cervical cancers after failure of cisplatin-based chemotherapy treatment or refusing chemotherapy. In this study, we will generate dendritic cells by culturing patient's autologous PBMC with GM-CSF and IL-4 in vitro. These dendritic cells will be pulsed with synthetic peptides representing the CTL epitopes on HPV Type 16 E7. Antigen-pulsed dendritic cells will be injected into inguinal lymph nodes under the guidance of real-time sonography. Each patient will receive four injections and 12 patients in total will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. recurrent cervical cancer
2. HPV 16 infection
3. Previously received cisplatin ot 5-FU based chemotherapy or refused to receive chemotherapy
4. HLA-A2 haplotype
5. Older than 20 years old
6. ECOG I or II
7. Life expectancy longer than 3 months
8. Adequate bone marrow reserve
9. pregnancy test: negative
10. Informed consent obtained

Exclusion Criteria:

1. CNS metastasis
2. Acute or chronic infection
3. Pregnant or lactating women
4. Asthma
5. Cardiac diseases such as heart failure, unstable angina, arrhythmia, myocardial infarction
6. Autoimmune disease
7. Previously other cancers (except basal cell cancer)
8. Without chemotherapy, biotherapy for more than 6 weeks

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2003-01; Study Completion 2006-03

PRIMARY OUTCOMES:
1. Safety issues in patients receiving HPV16 E7 peptide-pulsed autologous DCs immunotherapy

SECONDARY OUTCOMES:
1. Immunologic responses in patients receiving HPV16 E7 peptide-pulsed autologous DCs immunotherapy
2. Clinical response in patients receiving HPV16 E7 peptide-pulsed autologous DCs immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan